CLINICAL TRIAL: NCT06308120
Title: A Randomized Controlled Trial to Compare Robotic Assisted Bronchoscopy Ion's Clinical Utility for Peripheral Lung Nodule Access and Diagnosis to ENB
Brief Title: A Trial to Compare Robotic Assisted Bronchoscopy Ion's Clinical Utility for Peripheral Lung Nodule Access and Diagnosis to ENB
Acronym: ARTICULAtE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Collaborators: Intuitive Surgical-Fosun Medical Technology (Shanghai) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ISI-IONCN-002
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Nodule, Solitary; Lung Cancer
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Stratified, randomized controlled trial with parallel group assignment
Who Masked: Outcomes Assessor
Masking Description: Pathologist reviewing biopsy results will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ION™ Endoluminal System (Active Comparator): ION™ Endoluminal System Providers will utilize the ION™ Endoluminal System to perform a diagnostic bronchoscopy procedure
  Interventions: Device: Ion Endoluminal System
- superDimension Navigation System and Accessories (Active Comparator): Providers will utilize the superDimension Navigation System and Accessories to perform a diagnostic bronchoscopy procedure.
  Interventions: Device: superDimension Navigation System and Accessories

INTERVENTIONS:
Device: Ion Endoluminal System — Participants in the test arm will undergo a diagnostic bronchoscopy with ION™ Endoluminal System.
  Arms: ION™ Endoluminal System
Device: superDimension Navigation System and Accessories — Participants in the control arm will undergo a diagnostic bronchoscopy with superDimension Navigation System and Accessories.
  Arms: superDimension Navigation System and Accessories

SUMMARY:
Multi-center randomized controlled study designed to compare the diagnostic yield of ION™ Endoluminal System with electromagnetic navigation bronchoscopy in patients undergoing transbronchial sampling procedure of peripheral pulmonary nodules.

DETAILED DESCRIPTION:
Lung cancer is the malignant tumor with the highest morbidity and mortality in the world. Besides the aggressive nature of lung cancer, the overall high cancer mortality is mainly associated with the time delay between cancer development and initial clinical symptoms.

In the past, bronchoscope was mainly used to biopsy the nodules in the central airway but played a limited role in managing peripheral nodules due to its low diagnosis accuracy in such nodules. Advanced bronchoscopic techniques include tools for bronchoscopic guidance such as guide sheath (GS), Endobronchial Ultrasound (EBUS), Electromagnetic Navigation (ENB), or Virtual Bronchoscopic Navigation (VBN). In well-designed clinical studies, these techniques can be used to increase the diagnostic yield of flexible bronchoscope in dealing with peripheral nodules. However, the real-world registry study data showed that the diagnostic yield of these techniques in practice is as low as 53.7 %.. More importantly, these advanced bronchoscopic techniques haven't been widely used or become standard treatments in China mainly due to high skill requirements and high costs.

ION™ Endoluminal System is a robotic-assisted system which assists the user in navigating a catheter and endoscopic tools in the pulmonary tract under bronchial endoscope for diagnostic and therapeutic procedures. The fully articulating catheter with a small outer diameter of 3.5 mm can enter the small airways around the lungs with navigation enabled by shape-sensing technology and not electromagnetics; the shape sensing fiber provides instant feedbacks on shapes and locations during navigation and biopsy. The tool channel with an inner diameter of 2 mm for the catheter is compatible with various biopsy tools.

The purpose of this study a randomized controlled study to test the hypothesis that the diagnostic yield of ION™ is Superior to electromagnetic navigation bronchoscopy in patients undergoing bronchoscopy to biopsy a peripheral pulmonary nodule (PPN).

ELIGIBILITY:
Inclusion Criteria:

1. Able to tolerate bronchoscopy;
2. ≥18 years and ≤ 80 years;
3. Chest CT scan results suggest one or more pulmonary nodules and suspected pulmonary malignant tumor which requires further diagnostic evaluation*;
4. The pulmonary nodules are solid or part-solid;
5. The maximum diameter of the whole nodule is >8 mm and ≤30 mm;
6. Chest CT scan results suggest peripheral nodules which are defined as nodules in the Generation 4 or above of the airway (trachea is defined as Generation 0, left and right principal bronchi as Generation 1, lobar bronchi as Generation 2, segmental bronchi as Generation 3, and subsegmental bronchi as Generation 4);
7. Able to understand and adhere to study requirements;
8. Able to provide and sign the informed consent form.

Exclusion Criteria:

1. The target nodule has been diagnosed as a malignant tumor or metastatic tumor;
2. The target nodule is later determined as a central lesion (the target nodule is in the airway, and not at a subsegmental or more distal location) during the bronchoscopy before the study procedure starts;
3. Contraindications to bronchoscopy;
4. Contraindication to intubation, general anesthesia, or over American Society of Anesthesiologists (ASA) score of 3;
5. Known allergies, sensitivities, or previous allergic reactions to the disinfection reagents for reprocessing of the investigational product;
6. Pregnancy;
7. Any other condition that may increase the risk of bronchoscopic procedure as identified in the evaluation by the PI or bronchoscopist before bronchoscopic procedure;
8. Other conditions that the investigators consider not suitable for the subjects to participate in the study;
9. Participation in any other interventional or investigational clinical studies within 30 days before enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | 6 months post-procedure
  Diagnostic yield=number of study procedures in which a true positive for malignancy or a specific benign result is diagnosed by biopsy or non-specific benign is confirmed at the follow-up 6 months after procedure/total number of study procedures of each group ×100 %

SECONDARY OUTCOMES:
Sensitivity for malignancy of biopsy obtained samples | 6 months post-procedure
  Diagnostic sensitivity of malignancies=number of cases diagnosed with malignancies by study procedure / number of causes with malignancies in each group * 100 %
Incidence of pneumothorax that requires chest tube placement and/or re-hospitalization or extended hospitalization | 1 month post-procedure
  Pneumothorax is graded according to CTCAE 5.0. and differentiated according to the necessity to place a chest tube, readmission to the hospital, or prolonged hospitalization.
Incidence of intraoperative severe airway bleeding | Intra-procedure
  Severe airway bleeding is defined as Grade 3 or above per Nashville Delphi scale (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, M.D., Principal Investigator — Shanghai Chest Hospital
Locations (3):
- China (3):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu D, Li C, Xie F, Hu X, Shi J, Liu Z, Liu J, Simoff MJ, Song Y, Sun J. Shape-sensing robotic-assisted bronchoscopy (ss-RAB) for peripheral pulmonary nodules: learning curve and diagnostic performance from an initial multicenter experience in China. Respir Res. 2026 Jan 26. doi: 10.1186/s12931-025-03488-z. Online ahead of print. PMID 41588450
- [Derived] Xie F, Zhang C, Li C, Liu D, Song Y, Simoff MJ, Sun J. Protocol for robotic-assisted bronchoscopy versus electromagnetic navigation bronchoscopy for the diagnosis of peripheral pulmonary nodules: a randomized trial (ARTICULAtE study). J Thorac Dis. 2025 Jun 30;17(6):4339-4348. doi: 10.21037/jtd-2025-312. Epub 2025 Jun 26. PMID 40688277